CLINICAL TRIAL: NCT03128814
Title: The Degree, Development and Interrelationship of Structural and Functional Asymmetry in (Pre)Adolescent Elite Tennis Players: A Prospective Cohort Study With a Link to Growth and Maturation, Technical Skill Performance and Whole Body Injury
Brief Title: The Degree, Development and Interrelationship of Structural and Functional Asymmetry in (Pre)Adolescent Elite Tennis Players
Acronym: AsymTen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Laurent Chapelle (Other)
Responsible Party: Sponsor-Investigator, Laurent Chapelle, Researcher, Vrije Universiteit Brussel
Organization: Vrije Universiteit Brussel (Other)
Other Study IDs: Asymmetry in tennis
Record Dates: First submitted 2017-03-28; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Development; Unilateral
Keywords: Tennis; Asymmetry; Structural; Functional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elite (pre)adolescent tennis players
- Age- and gender-matched controls

SUMMARY:
Humans generally develop a preferred upper and lower extremity. Due to repetitive uneven loading, this gradually results in structural (e.g. increased bone and muscle mass) and functional (e.g. increased strength) adaptations to the dominant side of the body. The corresponding structural and functional asymmetry can be further accentuated by (intensively) practicing a unilateral sport such as tennis, which is very popular. Yet, research on this particular topic is scarce, especially in (pre)adolescent players. Existing studies, which often face methodological shortcomings (e.g. crosssectional designs, small sample sizes, no link to field methods), mainly focus on adults and structural asymmetry of the upper extremity itself, with very little or no attention to whole body structural as well as functional asymmetry. Moreover, the link of both forms of asymmetry with growth and maturation, everyday locomotion, technical skill performance and whole body injury is currently not (fully) understood. Therefore, the main purpose of this research project is to gain comprehensive knowledge on the degree, development and implications of both structural and functional asymmetry during a critical period in life using a longitudinal approach. As such, this project among youth elite tennis players will provide insights on the extent to which structural and/or functional asymmetry is acceptable for being most successful but remaining injury free.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in a Belgian high-performance tennis academy

Exclusion Criteria:

* Injury at the start of the data collection, any known musculoskeletal abnormality, developmental disorder or metabolic disease.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Young elite tennis players enrolled in Belgian high-performance tennis academies as well as age- and gender-matched (within two months) controls.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Anthropometry | September 2017 - December 2020
  Stature (cm) Sitting height (cm) Upper- and lower extremity length (cm) body weight (kg) Body Mass Index (kg/m²) Age at Peak height Velocity (years) Skeletal muscle mass (kg)
  These values will be determined every two months during a maximum period of three years, expressed as mean and standard deviation and will be used to develop growth charts and velocity curves.
Body composition | September 2017 - December 2020
  Dual X-Ray Absorptiometry
  * lean mass (g)
  * fat mass (g)
  * bone mass (g)
  * total bone area (cm²)
  * Bone Mineral Content (g)
  * Bone Mineral Density (g/cm²)
  Circumferences - upper and lower arm, thigh and calf (in cm)
  Ultrasound
  - Muscle thickness ((in mm) of M. Biceps, M. Triceps, M. Rectus Abdominis, Quadriceps and Hamstrings)
  Bioelectric impedance
  * fat (g)
  * fat free mass (g)
  These outcome measures will be determined on both the dominant and the non-dominant extremity/side every six months during a maximum period of three years. The side-to-side difference will be calculated using the symmetry index (see outcome measure 4). Every outcome measure described above will be expressed as mean and standard deviation for both the dominant and non-dominant extremity/side
Functional test battery | September 2017 - December 2020
  Strength and Power:
  * Seated shot put functional test (distance in cm)
  * Grip Strength (kg)
  * Unilateral countermovement jump (distance in cm)
  * Single hop test (distance in cm)
  * Medicine Ball throws (distance in cm)
  Speed and Agility:
  * Plate tapping (time s)
  * Single leg 6-m hop test (time in s)
  Balance and Flexibility:
  * Upper- and Lower extremity Y-balance test (distance in cm)
  * Standing On One Leg with Eyes Closed (time in s)
  Motor control and Coordination:
  * Unilateral hand wall toss test (score in points)
  * 270 degrees tap test (time in s)
  Locomotion pattern:
  - Ground Reaction Forces (force in N)
  Every test will be performed unilaterally for both the dominant and non-dominant extremity/side every six months during a maximum period of three years. The side-to-side difference will be calculated using the symmetry index (see outcome measure 4). The mean (plus standard deviation) of every test (dominant and non-dominant test score) will be reported
Structural and functional asymmetry index | September 2017 - December 2020
  Side-to-side difference (i.e. dominant vs non-dominant extremity/side) will be calculated and expressed as a percentage (extremity symmetry index (%)) for the outcome measures described above (anthropometry, body composition and functional test battery) using following formula:
  ((measure dominant extremity/measure non-dominant extremity)-1) x 100

SECONDARY OUTCOMES:
Injury incidence | September 2017 - December 2020
  Injury incidence in young elite tennis players (patterns and occurence) will be recorded and reported continuously for a maximum period of three years.
Technical tennis skills performance | September 2017 - December 2020
  technical skill of young elite tennis players. - Technical skill performance will be examined by means of video analysis once a year and scored by an independent expert panel. Mean technical ability will be reported.
  Tennis specific performance:
  - Tennis players will perform the Dutch Technical-Tactical Tennis Test (D4T) once a year. The mean test score will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Clarys, PhD, Study Director — Vrije Universiteit Brussel; Eva D'Hondt, PhD, Study Director — Vrije Universiteit Brussel
Locations (1):
- Physical Education and Physical Therapy, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared or will not be available to other researchers